CLINICAL TRIAL: NCT00393601
Title: Retrospective Chart Review of Laparoscopic Radical Cystectomy
Brief Title: Chart Review of Laparoscopic Radical Cystectomy
Status: Completed | Type: Observational
Sponsor: University of California, Irvine (Other)
Responsible Party: Atreya Dash, MD, University of California, Irvine
Other Study IDs: 2005-4596
Record Dates: First submitted 2006-10-27; First posted 2006-10-30 (Estimated); Last update posted 2010-01-06 (Estimated); Status verified 2010-01

CONDITIONS: Laparoscopic Radical Cystectomy
Keywords: Cystectomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigator intends to review retrospective de-identified data of patients who have had Laparoscopic Radical Cystectomies by the Department of Urology at UCIMC.

DETAILED DESCRIPTION:
The investigator fills out a standardized form for each patient undergoing a laparoscopic radical cystectomy.

ELIGIBILITY:
Inclusion Criteria:

* Review information on patients who had laparoscopic Radical cystectomy at UCIMC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Those who have undergone a laparoscopic radical cystectomy performed by Dr. David Ornstein.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2005-12; Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Atreya Dash, MD, Principal Investigator — University of California, Irvine
Locations (1):
- University of California, Irvine Medical Center, Orange, California, United States